CLINICAL TRIAL: NCT06088719
Title: Oncological Safety of Omitting Axillary Surgery in Breast Cancer Patients With Isolated Chest Wall Recurrence After Mastectomy
Brief Title: Safety of Omitting Axillary Surgery in Breast Cancer Patients With Isolated Chest Wall Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIRB Ref: 2019/2419
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Recurrent Disease
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- axillary surgery group: this group of patients had axillary surgery for axilla staging
  Interventions: Procedure: axillary surgery
- no axillary surgery group: this group of patients had no axillary surgery for axilla staging

INTERVENTIONS:
Procedure: axillary surgery — one group undergoes axillary surgery
  Groups: axillary surgery group

SUMMARY:
The axillary management of breast cancer patients with operable isolated chest wall recurrence after mastectomy is unclear. We aim to determine if axillary restaging surgery can be safely omitted with no increased recurrences in this group of patients.

ELIGIBILITY:
Inclusion Criteria: Mastectomy patients who developed pathologically confirmed invasive isolated chest wall recurrence.

-

Exclusion Criteria: -Patients with bilateral cancers

* Patients with evidence of concomitant distant or/and regional recurrences
* Patients who did not have surgery for their isolated chest wall recurrences.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with breast cancer with mastectomy and has isolated chest wall recurrences.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 1989-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence | from date of surgery to date of recurrence, up to 5 years
  axillary or distant recuurences

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore